CLINICAL TRIAL: NCT04892511
Title: A Randomized Trial on Hemodynamic Optimization of Cerebral Perfusion After Endovascular Therapy in Patients With Acute Ischemic Stroke (HOPE Study)
Brief Title: Hemodynamic Optimization of Cerebral Perfusion After Endovascular Therapy in Patients With Acute Ischemic Stroke
Acronym: HOPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-HOP-2021-01
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Labetalol; urapidil; Phenylephrine; Nitroprusside; Plasmalyte A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard treatment (No Intervention): Post-thrombectomy patients will have their blood pressure measured every hour for the first 24 hours after thrombectomy, and every 6 hours from 24 to 72 hours. The target blood pressure is not predefined by the study, but in patients who have received previous treatment with rt-PA, it is advisable to keep it below 180/110 mmHg. If the patient has not received rt-PA, there is no limitation, although the guidelines recommend keeping the pressure below 200/120 mmHg.
  The hypotensive or hypertensive treatments used will be noted.
- Optimized hemodynamic treatment (Experimental): Post-thrombectomy patients will have their blood pressure measured every 30 minutes for the first 24 hours after thrombectomy, and every 1 hour from 24 to 72 hours. Blood pressure objectives will depend on the degree of recanalization achieved after thrombectomy (see intervention section).
  The hypotensive or hypertensive treatments used will be noted.
  Interventions: Other: Adjusted medication

INTERVENTIONS:
Other: Adjusted medication — In patients randomized to perfusion optimization, medication will be adjusted to maintain blood pressure according to the degree of recanalization:
  * Patients with TICI 2b: systolic blood pressure 140-160 mmHg.
  * Patients with TICI 2c-3: systolic blood pressure <140 mmHg.
  Hypotensive drugs will be used when necessary. Intravenous labetalol is the treatment of choice, administered as a bolus or intravenous infusion. Alternative: urapidil (bolus or continuous infusion pump). If both drugs cannot be used or are insufficient, sodium nitroprusside can be used.
  Hypertensive drugs for TICI2b patients whose target pressure is 140-160mmHg and are below this range. Initially, a bolus of physiological saline or 100cc Plasmalyte® will be administered. If this treatment is not effective enough (blood pressure measurements persist <140 mmHg), intravenous phenylephrine will be administered.
  Other Names: Labetalol; Urapidil; Phenylephrine; Sodium Nitroprusside; Physiological saline or Plasmalyte®
  Arms: Optimized hemodynamic treatment

SUMMARY:
Mechanical thrombectomy is a very effective treatment in patients who have suffered an acute ischemic stroke associated with intracranial large vessel occlusion. However, less than half of the patients achieve functional independence despite treatment. The optimization of blood pressure after mechanical thrombectomy based on the degree of recanalization achieved at the end of the procedure could improve the perfusion of the ischemic brain tissue thanks to the improvement of blood circulation provided by collateral circulation. For this, authorized hypotensive or hypertensive drugs will be used. Moreover, this individualized treatment would allow to decrease reperfusion injury and therefore decrease the risk of intracerebral bleeding complications and cerebral edema. Therefore, we designed a clinical trial in which the standard management of blood pressure after mechanical thrombectomy will be compared with a specific protocol in which blood pressure targets are applied according to the degree of recanalization obtained during the thrombectomy procedure. The beneficial effect and risk reduction of this treatment will translate into a better short and long-term outcome

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ischemic stroke and large intracranial vessel occlusion within 24 hours after the onset of symptoms in whom mechanical thrombectomy has been performed.
* Successful recanalization, defined as a TICI score of 2b, 2c, or 3.
* Previous score on the modified Rankin scale (mRS) of 0, 1, or 2.
* The patient or her legal representative gives informed written or verbal consent

Exclusion Criteria:

* ASPECTS score <6
* Vertebral, basilar, A2, P2 and M3-4 occlusion
* History of intracerebral hemorrhage
* Pregnant or breastfeeding patient
* Patient with congestive heart failure or recent/unstable coronary artery disease (<3 months)
* Dissection of aorta, cervical or cerebral or unruptured aortic / cerebral aneurysm or known arteriovenous malformation
* Any bleeding visible on baseline CT
* History of ventricular arrhythmias
* Use of MAO inhibitors
* Inclusion in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 814 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale value | 3 months
  State of functional independence, measured with the modified Rankin scale at 3 months (+/- 14 days).

SECONDARY OUTCOMES:
NIHSS score | 24 hours
Mortality | 3 months
  Mortality from any cause at 3 months post-thrombectomy
Intracranial hemorrhagic complication | 24 hours
  Rate of any intracranial hemorrhagic complication in the first 24 hours after the procedure.
Intracranial hemorrhagic complication | 72 hours
  Rate of any intracranial hemorrhagic complication in the first 72 hours after the procedure.
Cerebral edema | 24 hours
  Volume of cerebral edema at 24 hours in the post-thrombectomy CT scan.
Cerebral edema | 72 hours
  Volume of cerebral edema at 72 hours in the post-thrombectomy CT scan.
Infarct size in the 24-hour post-thrombectomy CT. | 24 hours
  Infarct size in the 24-hour post-thrombectomy CT.
Infarct size in the 72-hour post-thrombectomy CT. | 72 hours
  Infarct size in the 72-hour post-thrombectomy CT.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Camps-Renom P, Guasch-Jimenez M, Martinez-Domeno A, Prats-Sanchez L, Ramos-Pachon A, Alvarez-Cienfuegos J, Silva Y, Fortea-Cabo G, Morales-Caba L, Rodriguez-Campello A, Giralt-Steinhauer E, Flores A, Ustrell X, Lopez-Hernandez N, Corona-Garcia DJ, Freijo-Guerrero MM, Luna A, Tejada-Meza H, Marta-Moreno J, Moniche F, Pardo-Galiana B, Castellanos M, Albert-Lacal L, Sanz-Monllor A, Aguilera-Simon A, Marin R, Ezcurra-Diaz G, Lambea-Gil A, Marti-Fabregas J. A Randomized Trial on Hemodynamic Optimization of Cerebral Perfusion after Successful Endovascular Therapy in Patients with Acute Ischemic Stroke (HOPE). Cerebrovasc Dis. 2025;54(4):559-566. doi: 10.1159/000540606. Epub 2024 Aug 29. PMID 39208776